CLINICAL TRIAL: NCT04289298
Title: Reaching and Engaging Depressed Senior Center Clients Phase II
Brief Title: Reaching and Engaging Depressed Senior Center Clients
Acronym: REDS II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-09020810-02; 5P50MH113838-03 (NIH)
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Depression in Old Age
Keywords: depression; geriatric; psychotherapy; group
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Engage-A (Experimental): Participants receive 9 individual in-person or remote therapy sessions. Each session will last approximately 60 minutes. During the sessions, the therapist will encourage the participant to engage in physical and social activities that are pleasurable or rewarding.
  Interventions: Behavioral: Engage-A
- Clinician (Experimental): Clinicians will be trained in Engage-A and supervised while utilizing the therapy.
  Interventions: Other: Training and utilizing Engage-A therapy

INTERVENTIONS:
Behavioral: Engage-A — Therapist will encourage participants to engage in physical and social activities that are pleasurable or rewarding. Engage is a stepped care psychotherapy based on what is known about how older adults respond to depression interventions. Stepped care is a model of treatment that starts with the minimum effective therapeutic techniques first, and then based on how well people respond to treatment, additional therapeutic techniques are added until people are recovered from their depression.
  Other Names: Augmented Engage
  Arms: Engage-A
Other: Training and utilizing Engage-A therapy — Therapist will be trained in Engage-A therapy and given supervision while utilizing this therapy.
  Arms: Clinician

SUMMARY:
The purpose of this study is to test the feasibility of one type of therapy session, Virtual Augmented Engage (Engage-A). The research is being done because the researchers are trying to learn if these approaches could be used by therapists in the community social service agencies to treat older adults with depression. The research will also measure clinician satisfaction after training and supervision of utilization of Engage-A.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years' old
* PHQ-9 Score of ≥ 10
* English or Spanish speaking
* MOCA ≥ 24 or mini-telephone MOCA ≥ 11
* Member of/attends one of the REDS Senior Centers
* Capacity to provide written consent for both research assessment and the Engage-A intervention.

Exclusion Criteria:

* Current active suicidal ideation defined by MADRS Suicide Item ≥ 4 (probably better off dead. Suicidal thoughts are common, and suicide is considered as a possible solution, but without specific plans or intention).
* Presence of psychiatric diagnoses other than unipolar, non-psychotic major depression or generalized anxiety disorder by SCID-IV.
* Severe or life-threatening medical illness (e.g., end stage organ failure).
* Currently seeing an individual psychotherapist *(if individuals are willing to go on a hiatus from their individual psychotherapist for the 15 weeks of the study, and meet all inclusion criteria, they will be considered eligible).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Marino, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this study is submitted to the National Database for Clinical Trials related to Mental Illness (NDCT). The NDCT is run by NIH and allows researchers studying mental health to collect and share information with each other. Researchers must apply to NIH in order to be allowed access to the data for 1 year's time; after which they must re-apply.
Time Frame: Data will be available as per NIMH's data sharing policy.
Access Criteria: Access criteria is determined by NIMH and can be requested by applying online.
URL: https://nda.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinician Participants: Clinicians who provided the ENGAGE intervention and participated in data collection about their experience.
Period: Overall Study
Arm/Group | Engage-A | Clinician Participants
Started | 22 | 4
Completed | 15 | 4
Not Completed | 7 | 0
Not completed — Lost to Follow-up | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engage-A | Clinician Participants | Total
Number analyzed (Participants) | 22 | 4 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.68 (6.53) | 48.5 (10.43) | 66.68 (6.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 4 | 24
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 19 | 2 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 18 | 4 | 22
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 4 | 26
Hamilton Psychiatric Rating Scale for Depression (HAM-D) [Mean (Standard Deviation); unit: units on a scale] — Hamilton Depression Rating Score (HAM-D) assesses the severity of depression in patients. The HAM-D ranges from 0 to 52, with higher scores indicating higher severity of depression. Population: The total number of ENGAGE-A participants analyzed differs from the overall total because 4 participants had incomplete baseline data.
  Depression scores were not collected for clinicians, as this measure is only appropriate for participants who are experiencing symptoms of depression.
  units on a scale
    number analyzed (Participants) | 18 | 0 | 18
    (all) | 21.28 (5.60) |  | 21.28 (5.60)
Behavioral Activation for Depression Scale (BADS) [Mean (Standard Deviation); unit: units on a scale] — The Behavioral Activation for Depression Scale (BADS) measures levels of behavioral activation. The BADS ranges from 0 to 150, with higher scores indicating lower levels of behavioral activation. Domain 1 scores range from 0-42. Higher scores (better outcome) indicate greater activation. Domain 2 scores range from 0-48. Higher scores (worse outcome) indicate greater Avoidance and Rumination. Domain 3 scores range from 0-30. Higher scores (worse outcome) indicate greater Work/School impairment. Domain 4 scores range from 0-30. Higher scores (worse outcome) indicate greater social impairment. Population: The number of ENGAGE-A participants analyzed for the baseline domains differs because two participants had incomplete responses for this questionnaire. The remaining rows differ due to participant withdrawal and loss to follow-up.
  Behavioral activation data were not collected for clinicians, as this measure is only appropriate for participants experiencing depressive symptoms.
  units on a scale
    Domain 1, Baseline: number analyzed (Participants) | 21 | 0 | 21
    Domain 1, Baseline | 18.62 (10.22) |  | 18.62 (10.22)
    Domain 2, Baseline: number analyzed (Participants) | 20 | 0 | 20
    Domain 2, Baseline | 22.50 (8.61) |  | 22.50 (8.61)
    Domain 3, Baseline: number analyzed (Participants) | 21 | 0 | 21
    Domain 3, Baseline | 13.76 (6.77) |  | 13.76 (6.77)
    Domain 4, Baseline: number analyzed (Participants) | 20 | 0 | 20
    Domain 4, Baseline | 20.25 (6.91) |  | 20.25 (6.91)

OUTCOME MEASURES:

1. Primary Outcome: Number of Virtual ENGAGE-A Participants Who Attend Every Scheduled Therapy Session
Description: Number of Virtual ENGAGE-A Participants who Attend Every Scheduled Therapy Session
Time Frame: 9 Weeks
Population: The total number of participants that completed all scheduled therapy sessions at week 9. The number of participants analyzed at week 9 for this measure (17) is higher than the number analyzed for the other measures at week 9 (16) because one participant attended the week 9 therapy session but left the study before having completed the week 9 assessment, during which the remaining measures are completed.
  Clinician Participants were not analyzed for this measure as it does not apply to them.
Measure: Count of Participants; unit: Participants
Arm/Group | Engage-A | Clinician Participants
Number analyzed (Participants) | 17 | 0
Participants | 17 |

2. Primary Outcome: Change in Average Satisfaction Score of Virtual ENGAGE-A Participants as Measured by the CSQ
Description: The Client Satisfaction Questionnaire (CSQ) assesses the clients' satisfaction with the services they are receiving. The CSQ ranges from 1-4, with higher scores indicating higher satisfaction. Domain 1 scores range from 1-4, with higher scores indicating higher satisfaction with the program. Domain 2 scores range from 1-4, with higher scores indicating higher satisfaction with the services received. Domain 3 scores range from 1-4, with higher scores indicating higher likelihood of wanting to receive similar services in the future. Higher scores for all three domains indicate a better outcome.
Time Frame: 6 weeks, 9 weeks, 12 weeks
Population: The number of participants analyzed at week 6 was 18, at week 9 was 16, and at week 12 was 15 due to loss to follow up and participant withdrawal.
  Clinician Participants were not analyzed for this measure as it does not apply to them.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engage-A | Clinician Participants
Number analyzed (Participants) | 18 | 0
units on a scale
  Domain 1- week 6 | 2.5 (0.62) |
  Domain 2- week 6 | 2.89 (0.76) |
  Domain 3- week 6 | 2.83 (0.79) |
  Domain 1- week 9: number analyzed (Participants) | 16 | 0
  Domain 1- week 9 | 2.5 (0.63) |
  Domain 2- week 9: number analyzed (Participants) | 16 | 0
  Domain 2- week 9 | 3.31 (0.79) |
  Domain 3- week 9: number analyzed (Participants) | 16 | 0
  Domain 3- week 9 | 3.33 (0.90) |
  Domain 1- week 12: number analyzed (Participants) | 15 | 0
  Domain 1- week 12 | 2.73 (0.88) |
  Domain 2- week 12: number analyzed (Participants) | 15 | 0
  Domain 2- week 12 | 3.40 (0.74) |
  Domain 3- week 12: number analyzed (Participants) | 15 | 0
  Domain 3- week 12 | 3.27 (0.88) |

3. Primary Outcome: Average Satisfaction Score of Community Clinicians (LCSW) as Measured by the TSQ
Description: The Therapist Satisfaction Questionnaire (TSQ) assesses the therapists' satisfaction with the Alacrity therapy training and intervention. The TSQ ranges from 1-4, with higher scores indicating higher satisfaction. Domain 1 scores range from 1-4, with higher scores indicating higher satisfaction with the skills obtained through training. Domain 2 scores range from 1-4, with higher scores indicating higher satisfaction with the therapy type. Domain 3 scores range from 1-4, with higher scores indicating higher likelihood that the therapist would use this therapy in their own practice. Higher scores for all three domains indicate better outcomes.
Time Frame: 2 years
Population: Engage-A participants were not analyzed as part of this measure as it does not apply to them.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Engage-A: Participants receive 9 individual in-person or remote therapy sessions. Each session will last approximately 60 minutes. During the sessions, the therapist will encourage the participant to engage in physical and social activities that are pleasurable or rewarding.
  Engage-A: Therapist will encourage participants to engage in physical and social activities that are pleasurable or rewarding. Engage is a stepped care psychotherapy based on what is known about how older adults respond to depression interventions. Stepped care is a model of treatment that starts with the minimum effective therapeutic techniques first, and then based on how well people respond to treatment, additional therapeutic techniques are added until people are recovered from their depression.
  Clinicians who provided the ENGAGE intervention and participated in data collection about their experience.
Arm/Group | Engage-A | Clinician Participants
Number analyzed (Participants) | 0 | 4
units on a scale
  Domain 1 |  | 4.0 (0.00)
  Domain 2 |  | 4.0 (0.00)
  Domain 3 |  | 4.0 (0.00)

4. Secondary Outcome: Change in Depressive Symptoms of Virtual ENGAGE-A Participants as Measured by HAM-D
Description: Hamilton Depression Rating Score (HAM-D) assesses the severity of depression in patients. The HAM-D ranges from 0 to 52, with higher scores indicating higher severity of depression.
Time Frame: Baseline, 6 week, 9 week, 12 week
Population: The total number of participants analyzed was 18 at baseline, 18 at week 6, 16 at week 9, and 15 and week 12 due to participant withdrawal and loss to follow-up.
  Clinician Participants were not analyzed for this measure as it does not apply to them.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engage-A | Clinician Participants
Number analyzed (Participants) | 18 | 0
units on a scale
  Baseline | 21.24 (5.77) |
  Week 6 | 14.47 (5.49) |
  Week 9: number analyzed (Participants) | 16 | 0
  Week 9 | 11.19 (5.65) |
  Week 12: number analyzed (Participants) | 15 | 0
  Week 12 | 11.67 (6.72) |

5. Secondary Outcome: Change in Behavioral Activation of Virtual ENGAGE-A Participants as Measured by the BADS
Description: The Behavioral Activation for Depression Scale (BADS) measures levels of behavioral activation.
  The BADS ranges from 0 to 150, with higher scores indicating lower levels of behavioral activation. Domain 1 scores range from 0-42. Higher scores (better outcome) indicate greater activation. Domain 2 scores range from 0-48. Higher scores (worse outcome) indicate greater Avoidance and Rumination. Domain 3 scores range from 0-30. Higher scores (worse outcome) indicate greater Work/School impairment. Domain 4 scores range from 0-30. Higher scores (worse outcome) indicate greater social impairment.
Time Frame: Baseline, 6 week, 9 week, 12 week
Population: The number of participants analyzed was 21 at baseline, 18 at week 6, 16 at week 9, and 15 at week 12.
  Clinician Participants were not analyzed for this measure as it does not apply to them.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engage-A | Clinician Participants
Number analyzed (Participants) | 21 | 0
units on a scale
  Domain 1, Baseline | 18.62 (10.22) |
  Domain 2, Baseline | 22.50 (8.61) |
  Domain 3, Baseline | 13.76 (6.77) |
  Domain 4, Baseline: number analyzed (Participants) | 18 | 0
  Domain 4, Baseline | 20.25 (6.91) |
  Domain 1, Week 6: number analyzed (Participants) | 18 | 0
  Domain 1, Week 6 | 24.67 (7.58) |
  Domain 2, Week 6: number analyzed (Participants) | 18 | 0
  Domain 2, Week 6 | 27.94 (8.77) |
  Domain 3, Week 6: number analyzed (Participants) | 18 | 0
  Domain 3, Week 6 | 16.61 (7.16) |
  Domain 4, Week 6: number analyzed (Participants) | 18 | 0
  Domain 4, Week 6 | 22.0 (7.23) |
  Domain 1, Week 9: number analyzed (Participants) | 16 | 0
  Domain 1, Week 9 | 27.94 (7.03) |
  Domain 2, Week 9: number analyzed (Participants) | 16 | 0
  Domain 2, Week 9 | 30.19 (11.23) |
  Domain 3, Week 9: number analyzed (Participants) | 16 | 0
  Domain 3, Week 9 | 20.19 (5.55) |
  Domain 4, Week 9: number analyzed (Participants) | 16 | 0
  Domain 4, Week 9 | 23.88 (5.89) |
  Domain 1, Week 12: number analyzed (Participants) | 15 | 0
  Domain 1, Week 12 | 24.40 (10.22) |
  Domain 2, Week 12: number analyzed (Participants) | 15 | 0
  Domain 2, Week 12 | 31.33 (12.83) |
  Domain 3, Week 12: number analyzed (Participants) | 15 | 0
  Domain 3, Week 12 | 21.47 (7.61) |
  Domain 4, Week 12: number analyzed (Participants) | 15 | 0
  Domain 4, Week 12 | 23.93 (8.24) |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 12 weeks for each Engage-A participant.
Description: Engage-A participants were assessed for adverse events. Clinicians were not assessed for adverse events.
Arm/Group | Engage-A | Clinician Participants
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/0
Other Adverse Events (participants affected / at risk) | 0/22 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT04289298/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT04289298/ICF_002.pdf